CLINICAL TRIAL: NCT05395741
Title: Evaluation of the Efficacy and Safety of Regorafenib in Patients With Refractory Primary Bone Tumors
Brief Title: Regorafenib in Patients With Refractory Primary Bone Tumors
Acronym: Regbone
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Institute of Mother and Child, Warsaw, Poland (Other)
Collaborators: Maria Sklodowska-Curie National Research Institute of Oncology (Other)
Responsible Party: Principal Investigator, Anna Raciborska, Head od Department of Oncology and Surgical Oncology for Children and Youth; Prof. Ass. PhD MD, Institute of Mother and Child, Warsaw, Poland
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Regbone
Record Dates: First submitted 2022-05-05; First posted 2022-05-27 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Osteosarcoma; Ewing Sarcoma of Bone
Keywords: TKI; refractory bone tumors; osteosarcoma; Ewing sarcoma; targeted treatment; solid tumor
MeSH Terms: conditions — Osteosarcoma; Bone Neoplasms; Sarcoma, Ewing | interventions — regorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- R1 - Regorafenib Arm (Experimental): R1 - the experimental group. Standard oncological treatment will be started. Additionally, patients will receive regorafenib orally at doses adjusted for age, body surface area and pharmacokinetics. Treatment with regorafenib will be continued for up to 1 year or until disease progression, patient death, unacceptable toxicity, or study closure. Pharmacokinetics and safety profile of the investigational product (IP) will be determined throughout the course therapy.
  Interventions: Drug: Regorafenib
- R2 - Control Group (No Intervention): R2 - the control group - will receive only standard treatment. In the event of progression or relapse, patients in the control group will have the option to receive the IP along with the standard treatment of the next line.

INTERVENTIONS:
Drug: Regorafenib — Patients will receive regorafenib orally at doses adjusted for age, body surface area and pharmacokinetics. Treatment with regorafenib will be continued for up to 1 year or until disease progression, patient death, unacceptable toxicity, or study closure. Pharmacokinetics and safety profile of the investigational product (IP) will be determined throughout the course therapy. In the event of progression or relapse, patients in the control group will have the option to receive the IP along with the standard treatment of the next line.
  Other Names: Stivarga
  Arms: R1 - Regorafenib Arm

SUMMARY:
The aim of the project is to improve treatment outcomes in patients with primary malignant bone tumors, refractory to standard therapy, by increasing the availability of advanced therapy, as well as to develop treatment options using advanced molecular diagnostics for patients who have not responded to the standard therapeutic regimen, and to introduce modern diagnostics for risk stratification and for the use in molecularly targeted therapies.

DETAILED DESCRIPTION:
The scope of the project is to cover the entire population of children, adolescents and young adults from the age of 9 to the age of 21, who progressed to first-line treatment or who presented with a recurrence of Ewing's sarcoma or osteosarcoma. Despite escalating doses of chemotherapy and radiotherapy, aggressive surgical procedures in patients with dissemination disease and negative prognostic factors, no improvement in treatment outcomes has been achieved for over 30 years. For this reason, other therapeutic options are being investigated. There have been no significant responses to immunotherapy. Although, the inclusion of tyrosine kinase inhibitors (TKIs) appears to be promising.

The identification of new mutations in bone tumors has led to a better insight into the molecular basis of these tumors, which has resulted in a more significant role of genetic research in everyday practice. Although traditional histopathological examinations are currently the basis for the diagnosis of bone tumors, the developing techniques of molecular biology make it possible, in many cases, to refine the diagnosis and, in the near future, will become the basis for the classification of these neoplasms. Moreover, these technics are expected to enable the qualification of patients to modern molecularly targeted therapies.

Based on the above data, the objectives of the project are as follows: 1. to estimate the nature and frequency of mutations in the tumor tissue, 2. to compare molecular test results with clinical data (which will allow for the initial assessment of the impact of the mutation status on the clinical condition, course of treatment and prognosis), 3. to include targeted treatment - broad spectrum tyrosine kinase inhibitor - regorafenib in standard therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Age >9 years ≤ 21 years.
2. Histologically proven Ewing sarcoma or osteosarcoma.
3. Failure of the treatment identified no earlier than 30 days prior to study treatment initiation (at least one of below needs to apply in order for this requirement to be satisfied):

   1. progression on the I line or next, or
   2. relapse.
4. Signing of informed consent for trial participation (including for Regorafenib treatment) according with current legal regulations.
5. Life expectancy of at least 12 weeks from the time informed consent was signed.
6. Possibility of swallowing the tablet.
7. Consent to the use of effective contraception throughout the period of the study and a minimum of 2 year after discontinuation of study treatment in patients at puberty and sexual maturity.

Exclusion Criteria:

1. Lack of inclusion criteria
2. Previous treatment with Regorafenib.
3. Pregnancy and breastfeeding.
4. Hypersensitivity to the study drug or any of its ingredients.
5. Simultaneous treatment with other drugs which might interact with Regorafenib.
6. Persistent toxicity related to prior therapy, making it impossible to treat with Regorafenib.
7. Diagnosis of other malignancies before study inclusion.
8. Patients with uncontrolled hypertension.
9. Patients with diseases of the coagulation system.
10. Patients with heart defects and / or cardiac arrhythmias requiring permanent treatment with antiarrhythmic drugs.
11. Other acute or persistent disorders, behaviors or abnormal laboratory test results, which might increase the risk related to the participation in this clinical trial or to taking the study drug, or which might influence the interpretation of the study results, or which, in the investigator's opinion, disqualify a patient from participating in the trial.

Ages: 9 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2022-04-28 (Actual); Primary Completion 2025-09-12 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
EFS - (Event-Free Survival). | 1 year
  To explore the efficacy in terms of EFS - (Event-Free Survival)
Determining the dose of the test substance in patients between 9 and 21 years of age, at which exposure to the drug will be similar to that recommended for adults. | 1 year
  Safety will be assessed by the rate of participants presenting with Adverse Events stratified by grade, category, affected organ or system, as number of serious adverse events (SAEs)
Assessment of safety in terms of AEs | from date of randomization, until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 48 months.
  Safety will be assessed by the rate of participants presenting with Adverse Events stratified by grade, category, affected organ or system, as number of adverse events (AEs), including adverse events of special interest
Assessment of the safety of regorafenib | from date of randomization, until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 48 months.
  Safety will be assessed by analyzing recorded vital signs, laboratory test results, echocardiography, and ECG.

SECONDARY OUTCOMES:
PFS (Progression-Free Survival). | Safety analyzes are planned in accordance with the schedule of intermediate analyzes, at least every 12 months.
  progression-free survival - will be measured from randomization to the detection of disease progression in imaging tests.
OS (Overall Survival). | Safety analyzes are planned in accordance with the schedule of intermediate analyzes, at least every 12 months.
  overall survival - will be measured from randomization to death due to cancer.
ORR (Overall Response Rate). | Safety analyzes are planned in accordance with the schedule of intermediate analyzes, at least every 12 months.
  the percentage of patients who achieved the response to treatment defined in the protocol.
Time to achieving sufficient drug concentration in serum. | Safety analyzes are planned in accordance with the schedule of intermediate analyzes, at least every 12 months.
  Concentration parameters will come directly from the concentration values measured in PK samples.
Maximum serum concentration in steady state Cmaxs. | Safety analyzes are planned in accordance with the schedule of intermediate analyzes, at least every 12 months.
  Concentration parameters will come directly from the concentration values measured in PK samples.
Minimum serum concentration in steady state Cminss. | Safety analyzes are planned in accordance with the schedule of intermediate analyzes, at least every 12 months.
  Concentration parameters will come directly from the concentration values measured in PK samples.
Random serum concentration in steady state Css. | Safety analyzes are planned in accordance with the schedule of intermediate analyzes, at least every 12 months.
  Concentration parameters will come directly from the concentration values measured in PK samples.
Drug exposure Ctau. | Safety analyzes are planned in accordance with the schedule of intermediate analyzes, at least every 12 months.
  by monitoring the patient's clinical and molecular status
Time to achieving steady state drug concentration in serum. | Safety analyzes are planned in accordance with the schedule of intermediate analyzes, at least every 12 months.
  by monitoring the patient's clinical and molecular status

CONTACTS AND LOCATIONS:
Overall Officials: Anna Raciborska, Prof., Principal Investigator — the Institue of Mother and Child
Locations (2):
- Poland (2):
  - the Institute of Mother and Child, Warsaw
  - Maria Sklodowska-Curie National Research Institute of Oncology, Warsaw

REFERENCES:
- [Result] Agulnik M, Attia S. Growing Role of Regorafenib in the Treatment of Patients with Sarcoma. Target Oncol. 2018 Aug;13(4):417-422. doi: 10.1007/s11523-018-0575-0. PMID 29931504
- [Result] Allard M, Khoudour N, Rousseau B, Joly C, Costentin C, Blanchet B, Tournigand C, Hulin A. Simultaneous analysis of regorafenib and sorafenib and three of their metabolites in human plasma using LC-MS/MS. J Pharm Biomed Anal. 2017 Aug 5;142:42-48. doi: 10.1016/j.jpba.2017.04.053. Epub 2017 May 1. PMID 28494338
- [Result] Berry V, Basson L, Bogart E, Mir O, Blay JY, Italiano A, Bertucci F, Chevreau C, Clisant-Delaine S, Liegl-Antzager B, Tresch-Bruneel E, Wallet J, Taieb S, Decoupigny E, Le Cesne A, Brodowicz T, Penel N. REGOSARC: Regorafenib versus placebo in doxorubicin-refractory soft-tissue sarcoma-A quality-adjusted time without symptoms of progression or toxicity analysis. Cancer. 2017 Jun 15;123(12):2294-2302. doi: 10.1002/cncr.30661. Epub 2017 Mar 10. PMID 28295221
- [Result] Bruix J, Qin S, Merle P, Granito A, Huang YH, Bodoky G, Pracht M, Yokosuka O, Rosmorduc O, Breder V, Gerolami R, Masi G, Ross PJ, Song T, Bronowicki JP, Ollivier-Hourmand I, Kudo M, Cheng AL, Llovet JM, Finn RS, LeBerre MA, Baumhauer A, Meinhardt G, Han G; RESORCE Investigators. Regorafenib for patients with hepatocellular carcinoma who progressed on sorafenib treatment (RESORCE): a randomised, double-blind, placebo-controlled, phase 3 trial. Lancet. 2017 Jan 7;389(10064):56-66. doi: 10.1016/S0140-6736(16)32453-9. Epub 2016 Dec 6. PMID 27932229
- [Result] Cardoso E, Mercier T, Wagner AD, Homicsko K, Michielin O, Ellefsen-Lavoie K, Cagnon L, Diezi M, Buclin T, Widmer N, Csajka C, Decosterd L. Quantification of the next-generation oral anti-tumor drugs dabrafenib, trametinib, vemurafenib, cobimetinib, pazopanib, regorafenib and two metabolites in human plasma by liquid chromatography-tandem mass spectrometry. J Chromatogr B Analyt Technol Biomed Life Sci. 2018 Apr 15;1083:124-136. doi: 10.1016/j.jchromb.2018.02.008. Epub 2018 Feb 8. PMID 29544202
- [Result] Davis KL, Fox E, Merchant MS, Reid JM, Kudgus RA, Liu X, Minard CG, Voss S, Berg SL, Weigel BJ, Mackall CL. Nivolumab in children and young adults with relapsed or refractory solid tumours or lymphoma (ADVL1412): a multicentre, open-label, single-arm, phase 1-2 trial. Lancet Oncol. 2020 Apr;21(4):541-550. doi: 10.1016/S1470-2045(20)30023-1. Epub 2020 Mar 17. PMID 32192573
- [Result] Davis LE, Bolejack V, Ryan CW, Ganjoo KN, Loggers ET, Chawla S, Agulnik M, Livingston MB, Reed D, Keedy V, Rushing D, Okuno S, Reinke DK, Riedel RF, Attia S, Mascarenhas L, Maki RG. Randomized Double-Blind Phase II Study of Regorafenib in Patients With Metastatic Osteosarcoma. J Clin Oncol. 2019 Jun 1;37(16):1424-1431. doi: 10.1200/JCO.18.02374. Epub 2019 Apr 23. PMID 31013172
- [Result] Dirksen U, Brennan B, Le Deley MC, Cozic N, van den Berg H, Bhadri V, Brichard B, Claude L, Craft A, Amler S, Gaspar N, Gelderblom H, Goldsby R, Gorlick R, Grier HE, Guinbretiere JM, Hauser P, Hjorth L, Janeway K, Juergens H, Judson I, Krailo M, Kruseova J, Kuehne T, Ladenstein R, Lervat C, Lessnick SL, Lewis I, Linassier C, Marec-Berard P, Marina N, Morland B, Pacquement H, Paulussen M, Randall RL, Ranft A, Le Teuff G, Wheatley K, Whelan J, Womer R, Oberlin O, Hawkins DS; Euro-E.W.I.N.G. 99 and Ewing 2008 Investigators. High-Dose Chemotherapy Compared With Standard Chemotherapy and Lung Radiation in Ewing Sarcoma With Pulmonary Metastases: Results of the European Ewing Tumour Working Initiative of National Groups, 99 Trial and EWING 2008. J Clin Oncol. 2019 Dec 1;37(34):3192-3202. doi: 10.1200/JCO.19.00915. Epub 2019 Sep 25. PMID 31553693
- [Result] Duffaud F, Mir O, Boudou-Rouquette P, Piperno-Neumann S, Penel N, Bompas E, Delcambre C, Kalbacher E, Italiano A, Collard O, Chevreau C, Saada E, Isambert N, Delaye J, Schiffler C, Bouvier C, Vidal V, Chabaud S, Blay JY; French Sarcoma Group. Efficacy and safety of regorafenib in adult patients with metastatic osteosarcoma: a non-comparative, randomised, double-blind, placebo-controlled, phase 2 study. Lancet Oncol. 2019 Jan;20(1):120-133. doi: 10.1016/S1470-2045(18)30742-3. Epub 2018 Nov 23. PMID 30477937